CLINICAL TRIAL: NCT02276703
Title: Comparison of the Skin Conductance Values and Patient Pain Scores During Minor Procedures in the ICU
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Med-Storm Innovation (Unknown); Hopital Foch (Other)
Responsible Party: Principal Investigator, Elizabeth H. Sinz, Professor, Milton S. Hershey Medical Center
Other Study IDs: STUDY00000725
Record Dates: First submitted 2014-10-24; First posted 2014-10-28 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Skin Conductance Monitor — monitors skin conductance values
  Other Names: Algesimeter

SUMMARY:
Pain in hospitalized patients has received increasing attention, however due to its subjective nature, it has defied objective, quantitative measurements. If a patient is able to communicate, pain may be assessed using standardized sentences, visual analog scales (VAS) or plain numeric scales.

When a patient is unable to communicate, a method that would allow the caregiver to continuously monitor patients' pain and alert the provider that the patient may be in pain would be quite useful. The Pain Monitor uses a novel measurement technique of analyzing changes in skin conductance that can be used in patients who are unable to provide a subjective pain score. This study will compare the relationship between the measurements taken by the PainMonitor and pain scores given by communicative patients to evaluate the safety and efficacy of this monitor during planned, routine procedures.

DETAILED DESCRIPTION:
Although pain must be assessed to be treated, it has been challenging to obtain consistent, objective, and quantifiable measurements. The best methods currently available are subjective scales communicated by the patient such as standardized sentences, visual analog scales (VAS), or plain numeric scales.

When a patient is unable to communicate, methods used to monitor pain are inadequate. A device that provides an objective assessment of pain in these patients would alert the patient's caregivers that the patient may be in pain and analgesic treatment is indicated.

Various methods (Evans et al, 2013; Kantor, 2014; Isnardon, 2013) have been proposed to monitor patients' reactions to nociceptive stimulation such as:

* changes in heart rate or blood pressure
* changes in microcirculation
* pupillometry
* EEG
* Auditory or somatosensory evoked potentials

All of these methods have been found lacking, mostly due to a lack of specificity for pain. Pupillometry is not suitable for long periods of measurement and is sensitive to concomitant treatment (e.g. opioids).

Galvanometry has the potential to provide specific information related to pain in patients who are unable to communicate.

Since sweat glands are the only organs controlled solely by the sympathetic nervous system, there is a reasonable chance that the use of galvanometry can provide a reliable means of assessing pain. There are numerous papers on this topic; searching in PUBmed on the key words "pain" and "skin conductance" results in more than 250 papers (selected references are included in the list below). The PainMonitor system uses galvanometry to monitor changes in skin conductance responses per sec mirroring the number of bursts in the skin sympathetic nerves. This creates a warning for caregivers to assess the potential that the patient is in pain.

ELIGIBILITY:
Inclusion Criteria

* Patients between the ages of 18-89 years (inclusive), in an adult ICU
* Patients admitted to the ICU who are able to communicate their pain and anxiety using a VAS
* Patients must be cooperative and not agitated.
* Planned to have a potentially painful procedure

Exclusion Criteria:

* Diagnosed neuropathic disease
* Use of neostigmine within the past 3 hours
* Use of regional anesthesia at the extremity where the device electrodes are placed

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Intensive Care Unit (ICU) patients between the ages of 18-89 years (inclusive), that are scheduled to receive a painful procedure. We are requesting a total population of 120 to allow for withdrawals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity with a confidence interval | 1 year
  Sensitivity and specificity with a confidence interval > 80 % when skin conductance responses per sec are > 0.13 and VAS is equal to or greater than 30 mm. This end point will be reached by 100 patients with at least 10 discrete measurements for each patient.

CONTACTS AND LOCATIONS:
Locations (2):
- Hershey Medical Center, Hershey, Pennsylvania, United States
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No